CLINICAL TRIAL: NCT01737723
Title: Collecting Data for an Electroencephalograph Based Algorithm for Detection of Onset and Deterioration of Acute Ischemic Stroke by Comparison to NIHSS
Brief Title: Electroencephalograph for Detection of Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Neurokeeper Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: 2011-NK-1
Record Dates: First submitted 2012-11-27; First posted 2012-11-29 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Stroke
Keywords: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: Stroke patients
  Interventions: Device: Neurokeeper stroke detector

INTERVENTIONS:
Device: Neurokeeper stroke detector — Monitoring stroke patients

SUMMARY:
The purpose of this study is Collecting data for an Electroencephalograph based algorithm for detection of onset and deterioration of Acute Ischemic Stroke by Comparison to NIHSS.

DETAILED DESCRIPTION:
Inclusion criteria study population Age > 18 years old. Acute stroke symptoms onset within 120 hours of inclusion, and as proximate to event as possible.

Acute ischemic moderate or severe hemispheric stroke (assessed as 5 points or more by NIHSS) and including patients treated by t-PA

Exclusion criteria study population Primary intracranial hemorrhage on admission by CT. Significant movement disorder. Previous major hemispheric stroke. Local skull or skin affliction which prevents electrodes application. Any known condition which in the opinion of the investigator may interfere with the protocol implementation.

Inclusion criteria Control Population

Age > 18 years old.

Exclusion criteria Control Population Primary intracranial hemorrhage on admission by CT. Significant movement disorder. Previous major hemispheric stroke. Local skull or skin affliction which prevents electrodes application. Migraine Any known condition which in the opinion of the investigator may interfere with the protocol implementation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Acute stroke symptoms onset within 120 hours of inclusion, and as proximate to event as possible.
* Acute ischemic moderate or severe hemispheric stroke (assessed as 5 points or more by NIHSS) and including patients treated by t-PA

Exclusion Criteria:

* Primary intracranial hemorrhage on admission by CT.
* Significant movement disorder.
* Previous major hemispheric stroke.
* Local skull or skin affliction which prevents electrodes application.
* Any known condition which in the opinion of the investigator may interfere with the protocol implementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-08

PRIMARY OUTCOMES:
Detection of stroke
  EEG base algorithm system to detect and monitor changes in cerebral electrophysiological parameters as compared to clinical evaluation as assessed by NIHSS score.

SECONDARY OUTCOMES:
Correlation to severity of stroke
  Correlations between EEG + ERP changes and clinical status as assessed by NIHSS score.

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel